CLINICAL TRIAL: NCT00653224
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled, Parallel-group Study Evaluating the Efficacy and Impact on Health-related Quality of Life of Levocetirizine 5 mg Once Daily Given for 2 Weeks in Subjects 18 yr of Age and Older With Seasonal Allergic Rhinitis
Brief Title: A Study Evaluating the Efficacy and Impact on Health-related Quality of Life of Levocetirizine in Adults With Seasonal Allergic Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A00431
Record Dates: First submitted 2008-04-01; First posted 2008-04-04 (Estimated); Results first posted 2009-11-17 (Estimated); Last update posted 2011-08-31 (Estimated); Status verified 2009-12

CONDITIONS: Seasonal Allergic Rhinitis
Keywords: levocetirizine; Xyzal; Seasonal Allergic Rhinitis; total symptom score; quality of life
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — levocetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Matched placebo tablets
  Interventions: Drug: placebo
- LCTZ (Experimental): 5 mg tablet
  Interventions: Drug: levocetirizine dihydrochloride

INTERVENTIONS:
Drug: levocetirizine dihydrochloride — 5 mg daily (oral tablet) for 14 days
  Other Names: Xyzal
  Arms: LCTZ
Drug: placebo — 0 mg daily (matching oral tablet) for 14 days
  Arms: Placebo

SUMMARY:
The study objective is to investigate the efficacy of levocetirizine in reducing symptoms associated with seasonal allergic rhinitis and in improving rhinitis-related Quality of Life.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a history of SAR symptoms
* A positive skin prick test at least one grass allergen
* Moderate - severe SAR symptoms at baseline
* Women of childbearing potential must use a medically acceptable form of contraception
* 80% compliance on run in study medication and 80% compliance on completing the diary

Exclusion Criteria:

* The presence of any clinically significant comorbid disease which may interfere with the study assessments
* The presence of renal disease
* Pregnant or breastfeeding
* Subject is currently participating in another clinical trial
* Known hypersensitivity to piperazines or any of the excipients
* Intake of medications prohibited before the start of the trial
* Subjects who started or changed the dose of immunotherapy
* Rhinitis medicamentosa
* Subjects with a recent history (within the last 2 years) of drug or alcohol abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Actual)
Dates: Start 2008-04; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (38):
- United States (38):
  - Tucson, Arizona
  - Los Angeles, California
  - Sacramento, California
  - San Francisco, California
  - San Jose, California
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Miami, Florida
  - Atlanta, Georgia
  - Gainesville, Georgia
  - Lawrenceville, Georgia
  - Stockbridge, Georgia
  - Normal, Illinois
  - Louisville, Kentucky
  - Harvard, Massachusetts
  - North Dartmouth, Massachusetts
  - Novi, Michigan
  - Minneapolis, Minnesota
  - Berlin, New Jersey
  - Skillman, New Jersey
  - Verona, New Jersey
  - Rochester, New York
  - Asheville, North Carolina
  - Charlotte, North Carolina
  - Wilmington, North Carolina
  - Cincinnati, Ohio
  - Edmond, Oklahoma
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Pittsburgh, Pennsylvania
  - Upland, Pennsylvania
  - Lincoln, Rhode Island
  - Germantown, Tennessee
  - San Antonio, Texas
  - Salt Lake City, Utah
  - South Burlington, Vermont
  - Arlington, Virginia
  - Milwaukee, Wisconsin

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 580 patients has been recruited and randomized. Baseline Characteristics describe all randomized subjects. Out of the 580 randomized subjects (ITT population), 578 subjects have been treated at least once (Safety population).
Groups:
- Placebo: Matching oral placebo tablet daily for 14 days
- Levocetirizine: Levocetirizine (LCTZ) 5 mg tablet daily for 14 days
Period: Overall Study
Arm/Group | Placebo | Levocetirizine
Started | 293 | 287
Completed | 286 | 280
Not Completed | 7 | 7
Not completed — Adverse Event | 2 | 1
Not completed — Lack of Efficacy | 1 | 2
Not completed — Loss of efficacy | 1 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Other | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Levocetirizine | Total
Number analyzed (Participants) | 293 | 287 | 580
Age Continuous [Mean (Standard Deviation); unit: years] | 37.53 (11.68) | 38.73 (11.50) | 38.13 (11.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 182 | 169 | 351
  Male | 111 | 118 | 229
Region of Enrollment [Number; unit: participants]
  United States | 293 | 287 | 580

OUTCOME MEASURES:

1. Primary Outcome: Mean 24-hour Reflective Total 5 Symptoms Score (T5SS) Over the Total Treatment Period (14 Days)
Description: Total 5 Symptoms Score (T5SS) is the sum of rhinorrhea, sneezing, nasal congestion, itchy nose and itchy eyes scores. Each individual symptom was scored from 0 (none) to 3 (severe). Total score ranges from 0 to 15.
Time Frame: Over the total treatment period (14 days)
Population: Number of participants from the Intent to treat (ITT) population with available T5SS over the Total Treatment Period
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 292 | 285
points on a scale | 8.68 (3.44) | 7.87 (3.17)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis for the primary endpoint is expressed as follows: 'The mean 24-hr reflective T5SS over the total treatment period is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — If the p-value of this estimated difference is lower than 5% the mean T5SS is considered as different between the two treatment groups; ANCOVA on the mean of T5SS including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.89, 95% CI [-1.33 to -0.45] — The difference presented is 'Levocetirizine 5 mg - Placebo'

2. Secondary Outcome: Change From Baseline in Overall Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Score at Endpoint During the Two-week Treatment Period
Description: The RQLQ is a validated instrument composed of 28 questions covering 7 dimensions of health. Each question is scored on a scale of 0 to 6 (in which 0 = not troubled and 6 = extremely troubled), and the mean value for each health dimension is calculated. Overall health-related quality of life is expressed as the mean of the seven dimension scores and ranges from 0 to 6. Endpoint is defined as the last available postbaseline measurement during the two week treatment period.
Time Frame: Baseline and at endpoint of the 2 week treatment period
Population: Number of participants from the ITT population with available overall RQLQ score at Endpoint visit and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 285
points on a scale | -0.93 (1.12) | -1.31 (1.15)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in overall RQLQ score at endpoint visit is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — If the p-value of this estimated difference is lower than 5% the mean change from baseline in overall RQLQ score is considered as different between the two treatment groups; ANCOVA on the change from baseline in overall RQLQ score including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.34, 95% CI [-0.52 to -0.17] — The difference presented is 'Levocetirizine 5 mg - Placebo'

3. Secondary Outcome: Change From Baseline in Overall Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Score at Week 1
Description: The RQLQ is a validated instrument composed of 28 questions covering 7 dimensions of health. Each question is scored on a scale of 0 to 6 (in which 0 = not troubled and 6 = extremely troubled), and the mean value for each health dimension is calculated. Overall health-related quality of life is expressed as the mean of the seven dimension scores and ranges from 0 to 6.
Time Frame: Baseline and week 1
Population: Number of participants from the ITT population with available RQLQ overall score at Visit 3 (Week 1) and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 288 | 282
points on a scale | -0.60 (0.93) | -0.94 (1.09)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in overall RQLQ score at visit 3 (week 1) is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.31, 95% CI [-0.47 to -0.15] — The difference presented is 'Levocetirizine 5 mg - Placebo'

4. Secondary Outcome: Change From Baseline in Overall Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Score at Week 2
Description: as for outcome 3
Time Frame: Baseline and week 2
Population: Number of participants from the ITT population with available overall RQLQ score at Visit 4 (Week 2) and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 286 | 279
points on a scale | -0.95 (1.12) | -1.34 (1.15)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in overall RQLQ score at visit 4 (week 2) is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.34, 95% CI [-0.52 to -0.17] — The difference presented is 'Levocetirizine 5 mg - Placebo'

5. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Activities Score at Endpoint During the Two-week Treatment Period
Description: The RQLQ is a validated instrument composed of 28 questions covering 7 dimensions of health. Each question is scored on a scale of 0 to 6 (in which 0 = not troubled and 6 = extremely troubled), and the mean value for each health dimension is calculated. Endpoint is defined as the last available postbaseline measurement during the two week treatment period.
Time Frame: Baseline and at endpoint of the 2 week treatment period
Population: Number of participants from the ITT population with available RQLQ activities score at Endpoint visit and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 241 | 233
points on a scale | -1.28 (1.39) | -1.55 (1.48)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in RQLQ activities score at endpoint visit is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.042, ANCOVA — If the p-value of this estimated difference is lower than 5% the mean change from baseline in RQLQ activities score is considered as different between the two treatment groups; ANCOVA on the change from baseline in RQLQ activities score including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.25, 95% CI [-0.49 to -0.01] — The difference presented is 'Levocetirizine 5 mg - Placebo'

6. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Activities Score at Week 1
Description: The RQLQ is a validated instrument composed of 28 questions covering 7 dimensions of health. Each question is scored on a scale of 0 to 6 (in which 0 = not troubled and 6 = extremely troubled), and the mean value for each health dimension is calculated.
Time Frame: Baseline and week 1
Population: Number of participants from the ITT population with available RQLQ activities score at Visit 3 (Week 1) and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 231 | 243
points on a scale | -0.80 (1.19) | -1.13 (1.41)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in RQLQ activities score at visit 3 (week 1) is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.014, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.29, 95% CI [-0.52 to -0.06] — The difference presented is 'Levocetirizine 5 mg - Placebo'

7. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Activities Score at Week 2
Description: as for outcome 6
Time Frame: Baseline and week 2
Population: Number of participants from the ITT population with available RQLQ activities score at Visit 4 (Week 2) and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 235 | 229
points on a scale | -1.30 (1.40) | -1.58 (1.48)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in RQLQ activities score at visit 4 (week 2) is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.036, ANCOVA — [p-value comment as in outcome 5, analysis 1]; [statistical method as in outcome 5, analysis 1]; Mean Difference (Final Values) = -0.26, 95% CI [-0.51 to -0.02] — The difference presented is 'Levocetirizine 5 mg - Placebo'

8. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Sleep Score at Endpoint During the Two-week Treatment Period
Description: as for outcome 5
Time Frame: Baseline and at endpoint of the 2 week treatment period
Population: Number of participants from the ITT population with available RQLQ sleep score at Endpoint visit and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 285
points on a scale | -0.90 (1.38) | -1.19 (1.40)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in RQLQ sleep score at endpoint visit is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.010, ANCOVA — If the p-value of this estimated difference is lower than 5% the mean change from baseline in RQLQ sleep score is considered as different between the two treatment groups; ANCOVA on the change from baseline in RQLQ sleep score including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.27, 95% CI [-0.48 to -0.07] — The difference presented is 'Levocetirizine 5 mg - Placebo'

9. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Sleep Score at Week 1
Description: as for outcome 6
Time Frame: Baseline and week 1
Population: Number of participants from the ITT population with available RQLQ sleep score at Visit 3 (Week 1) and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 288 | 282
points on a scale | -0.59 (1.29) | -0.84 (1.32)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in RQLQ sleep score at visit 3 (week 1) is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.026, ANCOVA — [p-value comment as in outcome 8, analysis 1]; [statistical method as in outcome 8, analysis 1]; Mean Difference (Final Values) = -0.23, 95% CI [-0.43 to -0.03] — The difference presented is 'Levocetirizine 5 mg - Placebo'

10. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Sleep Score at Week 2
Description: as for outcome 6
Time Frame: Baseline and week 2
Population: Number of participants from the ITT population with available RQLQ sleep score at Visit 4 (Week 2) and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 286 | 279
points on a scale | -0.93 (1.37) | -1.20 (1.40)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in RQLQ sleep score at visit 4 (week 2) is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.018, ANCOVA — [p-value comment as in outcome 8, analysis 1]; [statistical method as in outcome 8, analysis 1]; Median Difference (Final Values) = -0.25, 95% CI [-0.45 to -0.04] — The difference presented is 'Levocetirizine 5 mg - Placebo'

11. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Non-nose/Eye Symptoms Score at Endpoint During the Two-week Treatment Period
Description: as for outcome 5
Time Frame: Baseline and at endpoint of the 2 week treatment period
Population: Number of participants from the ITT population with available RQLQ non-nose/eye symptoms score at Endpoint visit and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 284
points on a scale | -0.71 (1.24) | -1.05 (1.26)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as: 'The mean change from baseline in RQLQ non-nose/eye symptoms score at endpoint visit is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.002, ANCOVA — If the p-value of this estimated difference is lower than 5% the mean change from baseline in RQLQ non-nose/eye symptoms score is considered as different between the two treatment groups; ANCOVA on the change from baseline in RQLQ N-N/E symptoms score including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.29, 95% CI [-0.47 to -0.10] — The difference presented is 'Levocetirizine 5 mg - Placebo'

12. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Non-nose/Eye Symptoms Score at Week 1
Description: as for outcome 6
Time Frame: Baseline and week 1
Population: Number of participants from the ITT population with available RQLQ non-nose/eye symptoms score at Visit 3 (Week 1) and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 286 | 281
points on a scale | -0.42 (1.08) | -0.70 (1.14)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in RQLQ non-nose/eye symptoms score at visit 3 (week 1) is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.006, ANCOVA — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.24, 95% CI [-0.41 to -0.07] — The difference presented is 'Levocetirizine 5 mg - Placebo'

13. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Non-nose/Eye Symptoms Score at Week 2
Description: as for outcome 6
Time Frame: Baseline and week 2
Population: Number of participants from the ITT population with available RQLQ non-nose/eye symptoms score at Visit 4 (Week 2) and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 286 | 278
points on a scale | -0.73 (1.25) | -1.08 (1.26)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in RQLQ non-nose/eye symptoms score at visit 4 (week 2) is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.003, ANCOVA — [p-value comment as in outcome 11, analysis 1]; [statistical method as in outcome 11, analysis 1]; Mean Difference (Final Values) = -0.28, 95% CI [-0.47 to -0.10] — The difference presented is 'Levocetirizine 5 mg - Placebo'

14. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Practical Problems Score at Endpoint During the Two-week Treatment Period
Description: as for outcome 5
Time Frame: Baseline and at endpoint of the 2 week treatment period
Population: Number of participants from the ITT population with available RQLQ practical problems score at Endpoint visit and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 292 | 284
points on a scale | -1.22 (1.50) | -1.62 (1.40)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in RQLQ practical problems score at endpoint visit is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — If the p-value of this estimated difference is lower than 5% the mean change from baseline in RQLQ practical problems score is considered as different between the two treatment groups; ANCOVA on the change from baseline in RQLQ practical pbs. score including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.39, 95% CI [-0.61 to -0.18] — The difference presented is 'Levocetirizine 5 mg - Placebo'

15. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Practical Problems Score at Week 1
Description: as for outcome 6
Time Frame: Baseline and week 1
Population: Number of participants from the ITT population with available RQLQ practical problems score at Visit 3 (Week 1) and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 288 | 282
points on a scale | -0.76 (1.26) | -1.14 (1.41)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in RQLQ practical problems score at visit 3 (week 1) is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 14, analysis 1]; Mean Difference (Final Values) = -0.36, 95% CI [-0.57 to -0.16] — The difference presented is 'Levocetirizine 5 mg - Placebo'

16. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Practical Problems Score at Week 2
Description: as for outcome 6
Time Frame: Baseline and week 2
Population: Number of participants from the ITT population with available RQLQ practical problems score at Visit 4 (Week 2) and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 285 | 278
points on a scale | -1.24 (1.51) | -1.66 (1.38)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in RQLQ practical problems score at visit 4 (week 2) is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 14, analysis 1]; [statistical method as in outcome 14, analysis 1]; Mean Difference (Final Values) = -0.40, 95% CI [-0.61 to -0.18] — The difference presented is 'Levocetirizine 5 mg - Placebo'

17. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Nasal Symptoms Score at Endpoint During the Two-week Treatment Period
Description: as for outcome 5
Time Frame: Baseline and at endpoint of the 2 week treatment period
Population: Number of participants from the ITT population with available RQLQ nasal symptoms score at Endpoint visit and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 292 | 284
points on a scale | -1.05 (1.45) | -1.45 (1.33)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in RQLQ nasal symptoms score at endpoint visit is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — If the p-value of this estimated difference is lower than 5% the mean change from baseline in RQLQ nasal symptoms score is considered as different between the two treatment groups; ANCOVA on the change from baseline in RQLQ nasal symptoms score including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.38, 95% CI [-0.59 to -0.18] — The difference presented is 'Levocetirizine 5 mg - Placebo'

18. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Nasal Symptoms Score at Week 1
Description: as for outcome 6
Time Frame: Baseline and week 1
Population: Number of participants from the ITT population with available RQLQ nasal symptoms score at Visit 3 (Week 1) and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 288 | 282
points on a scale | -0.68 (1.25) | -1.05 (1.25)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in RQLQ nasal symptoms score at visit 3 (week 1) is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 17, analysis 1]; [statistical method as in outcome 17, analysis 1]; Mean Difference (Final Values) = -0.35, 95% CI [-0.55 to -0.16] — The difference presented is 'Levocetirizine 5 mg - Placebo'

19. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Nasal Symptoms Score at Week 2
Description: as for outcome 6
Time Frame: Baseline and week 2
Population: Number of participants from the ITT population with available RQLQ nasal symptoms score at Visit 4 (Week 2) and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 285 | 278
points on a scale | -1.08 (1.46) | -1.49 (1.31)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in RQLQ nasal symptoms score at visit 4 (week 2) is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 17, analysis 1]; [statistical method as in outcome 17, analysis 1]; Mean Difference (Final Values) = -0.38, 95% CI [-0.59 to -0.17] — The difference presented is 'Levocetirizine 5 mg - Placebo'

20. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Eye Symptoms Score at Endpoint During the Two-week Treatment Period
Description: as for outcome 5
Time Frame: Baseline and at endpoint of the 2 week treatment period
Population: Number of participants from the ITT population with available RQLQ eye symptoms score at Endpoint visit and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 285
points on a scale | -0.88 (1.40) | -1.36 (1.41)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in RQLQ eye symptoms score at endpoint visit is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — If the p-value of this estimated difference is lower than 5% the mean change from baseline in RQLQ eye symptoms score is considered as different between the two treatment groups; ANCOVA on the change from baseline in RQLQ eye symptoms score including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.42, 95% CI [-0.63 to -0.21] — The difference presented is 'Levocetirizine 5 mg - Placebo'

21. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Eye Symptoms Score at Week 1
Description: as for outcome 6
Time Frame: Baseline and week 1
Population: Number of participants from the ITT population with available RQLQ eye symptoms score at Visit 3 (Week 1) and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 287 | 281
points on a scale | -0.62 (1.27) | -1.04 (1.32)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in RQLQ eye symptoms score at visit 3 (week 1) is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 20, analysis 1]; [statistical method as in outcome 20, analysis 1]; Mean Difference (Final Values) = -0.37, 95% CI [-0.56 to -0.17] — The difference presented is 'Levocetirizine 5 mg - Placebo'

22. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Eye Symptoms Score at Week 2
Description: as for outcome 6
Time Frame: Baseline and week 2
Population: Number of participants from the ITT population with available RQLQ eye symptoms score at Visit 4 (Week 2) and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 286 | 279
points on a scale | -0.89 (1.41) | -1.40 (1.40)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in RQLQ eye symptoms score at visit 4 (week 2) is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 20, analysis 1]; [statistical method as in outcome 20, analysis 1]; Mean Difference (Final Values) = -0.42, 95% CI [-0.63 to -0.22] — The difference presented is 'Levocetirizine 5 mg - Placebo'

23. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Emotional Score at Endpoint During the Two-week Treatment Period
Description: as for outcome 5
Time Frame: Baseline and at endpoint of the 2 week treatment period
Population: Number of participants from the ITT population with available RQLQ emotional score at Endpoint visit and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 285
points on a scale | -0.80 (1.36) | -1.21 (1.37)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in RQLQ emotional score at endpoint visit is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — If the p-value of this estimated difference is lower than 5% the mean change from baseline in RQLQ emotional score is considered as different between the two treatment groups; ANCOVA on the change from baseline in RQLQ emotional score including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.33, 95% CI [-0.53 to -0.13] — The difference presented is 'Levocetirizine 5 mg - Placebo'

24. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Emotional Score at Week 1
Description: as for outcome 6
Time Frame: Baseline and week 1
Population: Number of participants from the ITT population with available RQLQ emotional score at Visit 3 (Week 1) and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 287 | 281
points on a scale | -0.51 (1.17) | -0.91 (1.29)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in RQLQ emotional score at visit 3 (week 1) is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 23, analysis 1]; [statistical method as in outcome 23, analysis 1]; Mean Difference (Final Values) = -0.34, 95% CI [-0.52 to -0.15] — The difference presented is 'Levocetirizine 5 mg - Placebo'

25. Secondary Outcome: Change From Baseline in Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Emotional Score at Week 2
Description: as for outcome 6
Time Frame: Baseline and week 2
Population: Number of participants from the ITT population with available RQLQ emotional score at Visit 4 (Week 2) and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 286 | 279
points on a scale | -0.82 (1.37) | -1.24 (1.35)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in RQLQ emotional score at visit 4 (week 2) is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 23, analysis 1]; [statistical method as in outcome 23, analysis 1]; Mean Difference (Final Values) = -0.34, 95% CI [-0.53 to -0.14] — The difference presented is 'Levocetirizine 5 mg - Placebo'

26. Secondary Outcome: Total 5 Symptoms Score (T5SS) Over the First Week
Description: Total 5 Symptoms Score (T5SS) is the sum of rhinorrhea, sneezing, nasal congestion, itchy nose and itchy eyes scores. Each individual symptom was scored from 0 (none) to 3 (severe). T5SS ranges from 0 to 15. An average over the first week is provided.
Time Frame: Over week 1
Population: Number of participants from the ITT population with available T5SS over Week 1
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 292 | 284
points on a scale | 9.04 (3.37) | 8.24 (3.21)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean T5SS over week 1 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA on the mean of T5SS including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.89, 95% CI [-1.32 to -0.45] — The difference presented is 'Levocetirizine 5 mg - Placebo'

27. Secondary Outcome: Total 5 Symptoms Score (T5SS) Over the Second Week
Description: Total 5 Symptoms Score (T5SS) is the sum of rhinorrhea, sneezing, nasal congestion, itchy nose and itchy eyes scores. Each individual symptom was scored from 0 (none) to 3 (severe). T5SS ranges from 0 to 15. An average over the second week of treatment is provided.
Time Frame: Over week 2
Population: Number of participants from the ITT population with available T5SS over Week 2
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 286 | 279
points on a scale | 8.20 (3.80) | 7.41 (3.50)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean T5SS over week 2 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; ANCOVA on the mean of T5SS including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.88, 95% CI [-1.39 to -0.36] — The difference presented is 'Levocetirizine 5 mg - Placebo'

28. Secondary Outcome: Total 4 Symptoms Score (T4SS) Over the First Week
Description: Total 4 Symptoms Score (T4SS) is the sum of rhinorrhea, sneezing, itchy nose and itchy eyes scores. Each individual symptom was scored from 0 (none) to 3 (severe). T4SS ranges from 0 to 12. An average over the first week of treatment is provided.
Time Frame: Over week 1
Population: Number of participants from the ITT population with available T4SS over Week 1
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 292 | 284
points on a scale | 7.07 (2.80) | 6.32 (2.65)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean T4SS over Week 1 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — If the p-value of this estimated difference is lower than 5% the mean T4SS is considered as different between the two treatment groups; ANCOVA on the Mean T4SS including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.84, 95% CI [-1.20 to -0.49] — The difference presented is 'Levocetirizine 5 mg - Placebo'

29. Secondary Outcome: Total 4 Symptoms Score (T4SS) Over the Second Week
Description: Total 4 Symptoms Score (T4SS) is the sum of rhinorrhea, sneezing, itchy nose and itchy eyes scores. Each individual symptom was scored from 0 (none) to 3 (severe). T4SS ranges from 0 to 12. An average over the second week of treatment is provided.
Time Frame: Over week 2
Population: Number of participants from the ITT population with available T4SS over Week 2
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 286 | 279
points on a scale | 6.39 (3.13) | 5.74 (2.83)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean T4SS over Week 2 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; ANCOVA on the Mean T4SS including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.76, 95% CI [-1.18 to -0.35] — The difference presented is 'Levocetirizine 5 mg - Placebo'

30. Secondary Outcome: Total 4 Symptoms Score (T4SS) Over the Total Treatment Period (14 Days)
Description: Total 4 Symptoms Score (T4SS) is the sum of rhinorrhea, sneezing, itchy nose and itchy eyes scores. Each individual symptom was scored from 0 (none) to 3 (severe). T4SS ranges from 0 to 12. An average over the total treatment period of 14 days is provided.
Time Frame: Over total treatment period (14 days)
Population: Number of participants from the ITT population with available T4SS over the Total Treatment period
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 292 | 285
points on a scale | 6.78 (2.84) | 6.07 (2.59)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean T4SS over the total treatment period is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 28, analysis 1]; ANCOVA on the Mean T4SS including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.81, 95% CI [-1.17 to -0.45] — The difference presented is 'Levocetirizine 5 mg - Placebo'

31. Secondary Outcome: Total Nasal Symptom Score (TNSS) Over the First Week
Description: Total Nasal Symptoms Score (TNSS) is the sum of sneezing, rhinorrhea, nasal itching, nasal congestion and post-nasal drip scores. Each individual symptom was scored from 0 (none) to 3 (severe). TNSS ranges from 0 to 15. An average over the first week of treatment is provided.
Time Frame: Over week 1
Population: Number of participants from the ITT population with available TNSS over Week 1
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 292 | 285
points on a scale | 9.11 (3.39) | 8.34 (3.17)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean TNSS over Week 1 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — If the p-value of this estimated difference is lower than 5% the mean TNSS is considered as different between the two treatment groups; ANCOVA on the Mean TNSS including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.74, 95% CI [-1.17 to -0.31] — The difference presented is 'Levocetirizine 5 mg - Placebo'

32. Secondary Outcome: Total Nasal Symptom Score (TNSS) Over the Second Week
Description: Total Nasal Symptoms Score (TNSS) is the sum of sneezing, rhinorrhea, nasal itching, nasal congestion and post-nasal drip scores. Each individual symptom was scored from 0 (none) to 3 (severe). TNSS ranges from 0 to 15. An average over the second week of treatment is provided.
Time Frame: Over week 2
Population: Number of participants from the ITT population with available TNSS over Week 2
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 285 | 280
points on a scale | 8.23 (3.82) | 7.45 (3.52)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean TNSS over Week 2 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.005, ANCOVA — [p-value comment as in outcome 31, analysis 1]; ANCOVA on the Mean TNSS including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.74, 95% CI [-1.26 to -0.22] — The difference presented is 'Levocetirizine 5 mg - Placebo'

33. Secondary Outcome: Total Nasal Symptom Score (TNSS) Over the Total Treatment Period (14 Days)
Description: Total Nasal Symptoms Score (TNSS) is the sum of sneezing, rhinorrhea, nasal itching, nasal congestion and post-nasal drip scores. Each individual symptom was scored from 0 (none) to 3 (severe). TNSS ranges from 0 to 15. An average over the total treatment period is provided.
Time Frame: Over total treatment period (14 days)
Population: Number of participants from the ITT population with available TNSS over the Total Treatment period
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 292 | 285
points on a scale | 8.73 (3.45) | 7.94 (3.14)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean TNSS over the total treatment period is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 31, analysis 1]; ANCOVA on the Mean TNSS including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.74, 95% CI [-1.18 to -0.30] — The difference presented is 'Levocetirizine 5 mg - Placebo'

34. Secondary Outcome: Total Ocular Symptom Score (TOSS) Over the First Week
Description: Total Ocular Symptoms Score (TOSS) is the sum of ocular itching/burning, ocular tearing/watering and ocular redness scores. Each individual symptom was scored from 0 (none) to 3 (severe). TOSS ranges from 0 to 9. An average over the first week of treatment is provided.
Time Frame: Over week 1
Population: Number of participants from the ITT population with available TOSS over Week 1
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 285
points on a scale | 4.29 (2.54) | 3.99 (2.44)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean TOSS over Week 1 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — If the p-value of this estimated difference is lower than 5% the mean TOSS is considered as different between the two treatment groups; ANCOVA on the Mean TOSS including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.59, 95% CI [-0.87 to -0.30] — The difference presented is 'Levocetirizine 5 mg - Placebo'

35. Secondary Outcome: Total Ocular Symptom Score (TOSS) Over the Second Week
Description: Total Ocular Symptoms Score (TOSS) is the sum of ocular itching/burning, ocular tearing/watering and ocular redness scores. Each individual symptom was scored from 0 (none) to 3 (severe). TOSS ranges from 0 to 9. An average over the second week of treatment is provided.
Time Frame: Over week 2
Population: Number of participants from the ITT population with available TOSS over Week 2
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 285 | 280
points on a scale | 3.89 (2.64) | 3.60 (2.50)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean TOSS over Week 2 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 34, analysis 1]; ANCOVA on the Mean TOSS including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.57, 95% CI [-0.91 to -0.24] — The difference presented is 'Levocetirizine 5 mg - Placebo'

36. Secondary Outcome: Total Ocular Symptom Score (TOSS) Over the Total Treatment Period (14 Days)
Description: Total Ocular Symptoms Score (TOSS) is the sum of ocular itching/burning, ocular tearing/watering and ocular redness scores. Each individual symptom was scored from 0 (none) to 3 (severe). TOSS ranges from 0 to 9. An average over the total treatment period is provided.
Time Frame: Over total treatment period (14 days)
Population: Number of participants from the ITT population with available TOSS over the Total Treatment period
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 285
points on a scale | 4.13 (2.51) | 3.82 (2.39)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean TOSS over the total treatment period is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 34, analysis 1]; ANCOVA on the Mean TOSS including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.57, 95% CI [-0.86 to -0.28] — The difference presented is 'Levocetirizine 5 mg - Placebo'

37. Secondary Outcome: Sneezing Score Over the First Week
Description: The sneezing score ranges from 0 (none) to 3 (severe). An average over the first week of treatment is provided.
Time Frame: Over week 1
Population: Number of participants from the ITT population with available sneezing score over Week 1
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 292 | 285
points on a scale | 1.80 (0.82) | 1.57 (0.76)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The sneezing mean score over Week 1 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — If the p-value of this estimated difference is lower than 5% the sneezing mean score is considered as different between the two treatment groups; ANCOVA on the Sneezing Mean Score including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.23, 95% CI [-0.34 to -0.13] — The difference presented is 'Levocetirizine 5 mg - Placebo'

38. Secondary Outcome: Sneezing Score Over the Second Week
Description: The sneezing score ranges from 0 (none) to 3 (severe). An average over the second week of treatment is provided.
Time Frame: Over week 2
Population: Number of participants from the ITT population with available sneezing score over Week 2
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 286 | 280
points on a scale | 1.62 (0.88) | 1.41 (0.82)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The sneezing mean score over week 2 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 37, analysis 1]; ANCOVA on the Sneezing Mean Score including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.22, 95% CI [-0.34 to -0.09] — The difference presented is 'Levocetirizine 5 mg - Placebo'

39. Secondary Outcome: Sneezing Score Over the Total Treatment Period (14 Days)
Description: The sneezing score ranges from 0 (none) to 3 (severe). An average over the total treatment period is provided.
Time Frame: Over total treatment period (14 days)
Population: Number of participants from the ITT population with available sneezing score over the Total Treatment period
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 292 | 285
points on a scale | 1.72 (0.80) | 1.50 (0.73)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The sneezing mean score over the total treatment period is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 37, analysis 1]; ANCOVA on the Sneezing Mean Score including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.23, 95% CI [-0.33 to -0.12] — The difference presented is 'Levocetirizine 5 mg - Placebo'

40. Secondary Outcome: Rhinorrhea Score Over the First Week
Description: The rhinorrhea score ranges from 0 (none) to 3 (severe). An average over the first week of treatment is provided.
Time Frame: Over week 1
Population: Number of participants from the ITT population with available rhinorrhea score over Week 1
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 285
points on a scale | 1.81 (0.79) | 1.59 (0.79)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The rhinorrhea mean score over Week 1 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — If the p-value of this estimated difference is lower than 5% the rhinorrhea mean score is considered as different between the two treatment groups; ANCOVA on the Rhinorrhea Mean Score including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.21, 95% CI [-0.32 to -0.11] — The difference presented is 'Levocetirizine 5 mg - Placebo'

41. Secondary Outcome: Rhinorrhea Score Over the Second Week
Description: The rhinorrhea score ranges from 0 (none) to 3 (severe). An average over the second week of treatment is provided.
Time Frame: Over week 2
Population: Number of participants from the ITT population with available rhinorrhea score over Week 2
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 286 | 280
points on a scale | 1.63 (0.91) | 1.44 (0.84)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The rhinorrhea mean score over week 2 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.008, ANCOVA — [p-value comment as in outcome 40, analysis 1]; [statistical method as in outcome 40, analysis 1]; Mean Difference (Final Values) = -0.17, 95% CI [-0.30 to -0.05] — The difference presented is 'Levocetirizine 5 mg - Placebo'

42. Secondary Outcome: Rhinorrhea Score Over the Total Treatment Period (14 Days)
Description: The rhinorrhea score ranges from 0 (none) to 3 (severe). An average over the total treatment period is provided.
Time Frame: Over total treatment period (14 days)
Population: Number of participants from the ITT population with available rhinorrhea score over the Total Treatment period
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 285
points on a scale | 1.73 (0.80) | 1.53 (0.76)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The rhinorrhea mean score over the total treatment period is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 40, analysis 1]; [statistical method as in outcome 40, analysis 1]; Mean Difference (Final Values) = -0.19, 95% CI [-0.30 to -0.09] — The difference presented is 'Levocetirizine 5 mg - Placebo'

43. Secondary Outcome: Nasal Congestion Score Over the First Week
Description: The nasal congestion score ranges from 0 (none) to 3 (severe). An average over the first week of treatment is provided.
Time Frame: Over week 1
Population: Number of participants from the ITT population with available nasal congestion score over Week 1
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 285
points on a scale | 1.98 (0.78) | 1.92 (0.76)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The nasal congestion mean score over week 1 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.384, ANCOVA — If the p-value of this estimated difference is lower than 5% the nasal congestion mean score is considered as different between the two treatment groups; ANCOVA on the Nasal Congestion Mean Score including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.05, 95% CI [-0.15 to 0.06] — The difference presented is 'Levocetirizine 5 mg - Placebo'

44. Secondary Outcome: Nasal Congestion Score Over the Second Week
Description: The nasal congestion score ranges from 0 (none) to 3 (severe). An average over the second week of treatment is provided.
Time Frame: Over week 2
Population: Number of participants from the ITT population with available nasal congestion score over Week 2
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 286 | 280
points on a scale | 1.81 (0.89) | 1.67 (0.84)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The nasal congestion mean score over week 2 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.063, ANCOVA — [p-value comment as in outcome 43, analysis 1]; [statistical method as in outcome 43, analysis 1]; Mean Difference (Final Values) = -0.12, 95% CI [-0.24 to 0.01] — The difference presented is 'Levocetirizine 5 mg - Placebo'

45. Secondary Outcome: Nasal Congestion Score Over the Total Treatment Period (14 Days)
Description: The nasal congestion score ranges from 0 (none) to 3 (severe). An average over the total treatment period is provided.
Time Frame: Over total treatment period (14 days)
Population: Number of participants from the ITT population with available nasal congestion score over the Total Treatment period
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 285
points on a scale | 1.91 (0.79) | 1.80 (0.75)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The nasal congestion mean score over the total treatment period is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.124, ANCOVA — [p-value comment as in outcome 43, analysis 1]; [statistical method as in outcome 43, analysis 1]; Mean Difference (Final Values) = -0.08, 95% CI [-0.19 to 0.02] — The difference presented is 'Levocetirizine 5 mg - Placebo'

46. Secondary Outcome: Nasal Pruritus Score Over the First Week
Description: The nasal pruritus score ranges from 0 (none) to 3 (severe). An average over the first week of treatment is provided.
Time Frame: Over week 1
Population: Number of participants from the ITT population with available nasal pruritus score over Week 1
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 285
points on a scale | 1.80 (0.81) | 1.61 (0.79)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The nasal pruritus mean score over week 1 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.002, ANCOVA — If the p-value of this estimated difference is lower than 5% the nasal pruritus mean score is considered as different between the two treatment groups; ANCOVA on the Nasal Pruritus Mean Score including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.17, 95% CI [-0.28 to -0.06] — The difference presented is 'Levocetirizine 5 mg - Placebo'

47. Secondary Outcome: Nasal Pruritus Score Over the Second Week
Description: The nasal pruritus score ranges from 0 (none) to 3 (severe). An average over the second week of treatment is provided.
Time Frame: Over week 2
Population: Number of participants from the ITT population with available nasal pruritus score over Week 2
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 286 | 280
points on a scale | 1.63 (0.90) | 1.45 (0.84)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The nasal pruritus mean score over week 2 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.016, ANCOVA — [p-value comment as in outcome 46, analysis 1]; [statistical method as in outcome 46, analysis 1]; Mean Difference (Final Values) = -0.15, 95% CI [-0.28 to -0.03] — The difference presented is 'Levocetirizine 5 mg - Placebo'

48. Secondary Outcome: Nasal Pruritus Score Over the Total Treatment Period (14 Days)
Description: The nasal pruritus score ranges from 0 (none) to 3 (severe). An average over the total treatment period is provided.
Time Frame: Over total treatment period (14 days)
Population: Number of participants from the ITT population with available nasal pruritus score over the Total Treatment period
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 285
points on a scale | 1.73 (0.81) | 1.54 (0.76)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The nasal pruritus mean score over the total treatment period is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.003, ANCOVA — [p-value comment as in outcome 46, analysis 1]; [statistical method as in outcome 46, analysis 1]; Mean Difference (Final Values) = -0.16, 95% CI [-0.27 to -0.06] — The difference presented is 'Levocetirizine 5 mg - Placebo'

49. Secondary Outcome: Post-nasal Drip Score Over the First Week
Description: The post-nasal drip score ranges from 0 (none) to 3 (severe). An average over the first week of treatment is provided.
Time Frame: Over week 1
Population: Number of participants from the ITT population with available post-nasal drip score over Week 1
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 285
points on a scale | 1.72 (0.91) | 1.65 (0.87)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The post-nasal drip mean score over week 1 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.088, ANCOVA — If the p-value of this estimated difference is lower than 5% the post-nasal drip mean score is considered as different between the two treatment groups; ANCOVA on the Post-Nasal Drip Mean Score including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.09, 95% CI [-0.20 to 0.01] — The difference presented is 'Levocetirizine 5 mg - Placebo'

50. Secondary Outcome: Post-nasal Drip Score Over the Second Week
Description: The post-nasal drip score ranges from 0 (none) to 3 (severe). An average over the second week of treatment is provided.
Time Frame: Over week 2
Population: Number of participants from the ITT population with available post-nasal drip score over Week 2
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 285 | 280
points on a scale | 1.55 (0.99) | 1.48 (0.94)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The post-nasal drip mean score over Week 2 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.117, ANCOVA — [p-value comment as in outcome 49, analysis 1]; [statistical method as in outcome 49, analysis 1]; Mean Difference (Final Values) = -0.10, 95% CI [-0.23 to 0.03] — The difference presented is 'Levocetirizine 5 mg - Placebo'

51. Secondary Outcome: Post-nasal Drip Score Over the Total Treatment Period (14 Days)
Description: The post-nasal drip score ranges from 0 (none) to 3 (severe). An average over the total treatment period is provided.
Time Frame: Over total treatment period (14 days)
Population: Number of participants from the ITT population with available post-nasal drip score over the Total Treatment period
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 285
points on a scale | 1.64 (0.91) | 1.57 (0.85)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The post-nasal drip mean score over the total treatment period is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.065, ANCOVA — [p-value comment as in outcome 49, analysis 1]; [statistical method as in outcome 49, analysis 1]; Mean Difference (Final Values) = -0.10, 95% CI [-0.21 to 0.01] — The difference presented is 'Levocetirizine 5 mg - Placebo'

52. Secondary Outcome: Ocular Pruritus Score Over the First Week
Description: The ocular pruritus score ranges from 0 (none) to 3 (severe). An average over the first week of treatment is provided.
Time Frame: Over week 1
Population: Number of participants from the ITT population with available ocular pruritus score over Week 1
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 284
points on a scale | 1.65 (0.85) | 1.56 (0.82)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The ocular pruritus mean score over week 1 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — If the p-value of this estimated difference is lower than 5% the ocular pruritus mean score is considered as different between the two treatment groups; ANCOVA on the Ocular Pruritus Mean Score including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.21, 95% CI [-0.32 to -0.10] — The difference presented is 'Levocetirizine 5 mg - Placebo'

53. Secondary Outcome: Ocular Pruritus Score Over the Second Week
Description: The ocular pruritus score ranges from 0 (none) to 3 (severe). An average over the second week of treatment is provided.
Time Frame: Over week 2
Population: Number of participants from the ITT population with available ocular pruritus score over Week 2
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 286 | 279
points on a scale | 1.52 (0.92) | 1.44 (0.84)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The ocular pruritus mean score over week 2 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.002, ANCOVA — [p-value comment as in outcome 52, analysis 1]; [statistical method as in outcome 52, analysis 1]; Mean Difference (Final Values) = -0.20, 95% CI [-0.33 to -0.08] — The difference presented is 'Levocetirizine 5 mg - Placebo'

54. Secondary Outcome: Ocular Pruritus Score Over the Total Treatment Period (14 Days)
Description: The ocular pruritus score ranges from 0 (none) to 3 (severe). An average over the total treatment period is provided.
Time Frame: Over total treatment period (14 days)
Population: Number of participants from the ITT population with available ocular pruritus score over the Total Treatment period
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 285
points on a scale | 1.59 (0.84) | 1.51 (0.79)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The ocular pruritus mean score over the total treatment period is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 52, analysis 1]; [statistical method as in outcome 52, analysis 1]; Mean Difference (Final Values) = -0.21, 95% CI [-0.32 to -0.10] — The difference presented is 'Levocetirizine 5 mg - Placebo'

55. Secondary Outcome: Ocular Itching/Burning Score Over the First Week
Description: The ocular itching/burning score ranges from 0 (none) to 3 (severe). An average over the first week of treatment is provided.
Time Frame: Over week 1
Population: Number of participants from the ITT population with available ocular itching/burning score over Week 1
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 285
points on a scale | 1.58 (0.90) | 1.53 (0.86)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The ocular itching/burning mean score over Week 1 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — If the p-value of this estimated difference is lower than 5% the ocular itching/burning mean score is considered as different between the two treatment groups; ANCOVA on the Ocular Itching/Burning Mean Score including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.19, 95% CI [-0.30 to -0.08] — The difference presented is 'Levocetirizine 5 mg - Placebo'

56. Secondary Outcome: Ocular Itching/Burning Score Over the Second Week
Description: The ocular itching/burning score ranges from 0 (none) to 3 (severe). An average over the second week of treatment is provided.
Time Frame: Over week 2
Population: Number of participants from the ITT population with available ocular itching/burning score over Week 2
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 285 | 280
points on a scale | 1.42 (0.95) | 1.39 (0.90)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The ocular itching/burning mean score over Week 2 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.006, ANCOVA — [p-value comment as in outcome 55, analysis 1]; [statistical method as in outcome 55, analysis 1]; Mean Difference (Final Values) = -0.17, 95% CI [-0.29 to -0.05] — The difference presented is 'Levocetirizine 5 mg - Placebo'

57. Secondary Outcome: Ocular Itching/Burning Score Over the Total Treatment Period (14 Days)
Description: The ocular itching/burning score ranges from 0 (none) to 3 (severe). An average over the total treatment period is provided.
Time Frame: Over total treatment period (14 days)
Population: Number of participants from the ITT population with available ocular itching/burning score over the Total Treatment period
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 285
points on a scale | 1.52 (0.89) | 1.47 (0.84)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The ocular itching/burning mean score over the total treatment period is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 55, analysis 1]; [statistical method as in outcome 55, analysis 1]; Mean Difference (Final Values) = -0.18, 95% CI [-0.29 to -0.08] — The difference presented is 'Levocetirizine 5 mg - Placebo'

58. Secondary Outcome: Ocular Tearing/Watering Score Over the First Week
Description: The ocular tearing/watering score ranges from 0 (none) to 3 (severe). An average over the first week of treatment is provided.
Time Frame: Over week 1
Population: Number of participants from the ITT population with available ocular tearing/watering score over Week 1
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 285
points on a scale | 1.40 (0.91) | 1.26 (0.88)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The ocular tearing/watering mean score over week 1 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — If the p-value of this estimated difference is lower than 5% the ocular tearing/watering mean score is considered as different between the two treatment groups; ANCOVA on the Ocular Tearing/Watering Mean Score including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.20, 95% CI [-0.31 to -0.10] — The difference presented is 'Levocetirizine 5 mg - Placebo'

59. Secondary Outcome: Ocular Tearing/Watering Score Over the Second Week
Description: The ocular tearing/watering score ranges from 0 (none) to 3 (severe). An average over the second week of treatment is provided.
Time Frame: Over week 2
Population: Number of participants from the ITT population with available ocular tearing/watering score over Week 2
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 285 | 280
points on a scale | 1.27 (0.96) | 1.16 (0.91)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The ocular tearing/watering mean score over week 2 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.011, ANCOVA — [p-value comment as in outcome 58, analysis 1]; [statistical method as in outcome 58, analysis 1]; Mean Difference (Final Values) = -0.16, 95% CI [-0.29 to -0.04] — The difference presented is 'Levocetirizine 5 mg - Placebo'

60. Secondary Outcome: Ocular Tearing/Watering Score Over the Total Treatment Period (14 Days)
Description: The ocular tearing/watering score ranges from 0 (none) to 3 (severe). An average over the total treatment period is provided.
Time Frame: Over total treatment period (14 days)
Population: Number of participants from the ITT population with available ocular tearing/watering score over the Total Treatment period
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 285
points on a scale | 1.34 (0.89) | 1.22 (0.85)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The ocular tearing/watering mean score over the total treatment period is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 58, analysis 1]; [statistical method as in outcome 58, analysis 1]; Mean Difference (Final Values) = -0.18, 95% CI [-0.29 to -0.08] — The difference presented is 'Levocetirizine 5 mg - Placebo'

61. Secondary Outcome: Ocular Redness Score Over the First Week
Description: The ocular redness score ranges from 0 (none) to 3 (severe). An average over the first week of treatment is provided.
Time Frame: Over week 1
Population: Number of participants from the ITT population with available ocular redness score over Week 1
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 285
points on a scale | 1.31 (0.91) | 1.21 (0.93)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The ocular redness mean score over week 1 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.004, ANCOVA — If the p-value of this estimated difference is lower than 5% the ocular redness mean score is considered as different between the two treatment groups; ANCOVA on the Ocular Redness Mean Score including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.16, 95% CI [-0.27 to -0.05] — The difference presented is 'Levocetirizine 5 mg - Placebo'

62. Secondary Outcome: Ocular Redness Score Over the Second Week
Description: The ocular redness score ranges from 0 (none) to 3 (severe). An average over the second week of treatment is provided.
Time Frame: Over week 2
Population: Number of participants from the ITT population with available ocular redness score over Week 2
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 285 | 280
points on a scale | 1.20 (0.93) | 1.05 (0.93)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The ocular redness mean score over week 2 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 61, analysis 1]; [statistical method as in outcome 61, analysis 1]; Mean Difference (Final Values) = -0.22, 95% CI [-0.34 to -0.10] — The difference presented is 'Levocetirizine 5 mg - Placebo'

63. Secondary Outcome: Ocular Redness Score Over the Total Treatment Period (14 Days)
Description: The ocular redness score ranges from 0 (none) to 3 (severe). An average over the total treatment period is provided.
Time Frame: Over total treatment period (14 days)
Population: Number of participants from the ITT population with available ocular redness score over the Total Treatment period
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 285
points on a scale | 1.27 (0.89) | 1.14 (0.90)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The ocular redness mean score over the total treatment period is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 61, analysis 1]; [statistical method as in outcome 61, analysis 1]; Mean Difference (Final Values) = -0.19, 95% CI [-0.29 to -0.08] — The difference presented is 'Levocetirizine 5 mg - Placebo'

64. Secondary Outcome: Global Patient's Rating of Efficacy at Endpoint of the Two Week Treatment Period
Description: Endpoint is defined as the last available postbaseline measurement during the two week treatment period.Patient had to tick a box going from "Marked worsening" to "Marked improvement".
Time Frame: Baseline and at endpoint of the 2 week treatment period
Population: Number of participants from the ITT population
Measure: Number; unit: participants
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 287
participants
  Marked Worsening | 14 | 6
  Moderate Worsening | 16 | 11
  Slight Worsening | 21 | 8
  No Change | 86 | 69
  Slight Improvement | 81 | 95
  Moderate Improvement | 52 | 62
  Marked Improvement | 22 | 33
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Wilcoxon-Mann-Whitney, or Wilcoxon rank-sum test is generally used to detect 'shift alternatives'. That is, the two distributions have the same general shape, but one of them is shifted relative to the other by a constant amount under the alternative hypothesis; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — If the p-value is lower than 5% the distribution is considered as different between the two treatment groups

65. Secondary Outcome: Global Physician's Rating of Efficacy at Endpoint During the Two Week Treatment Period
Description: Endpoint is defined as the last available postbaseline measurement during the two week treatment period.Physician had to tick a box going from "Marked worsening" to "Marked improvement".
Time Frame: Baseline and at endpoint of the 2 week treatment period
Population: Number of participants from the ITT population
Measure: Number; unit: participants
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 287
participants
  Marked Worsening | 5 | 5
  Moderate Worsening | 13 | 7
  Slight Worsening | 18 | 7
  No Change | 106 | 70
  Slight Improvement | 75 | 92
  Moderate Improvement | 50 | 65
  Marked Improvement | 25 | 38
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Wilcoxon-Mann-Whitney, or Wilcoxon rank-sum test (Lehmann, 1975 page 23) is generally used to detect 'shift alternatives'. That is, the two distributions have the same general shape, but one of them is shifted relative to the other by a constant amount under the alternative hypothesis; Test type: Superiority or Other; p < 0.001, Wilcoxon (Mann-Whitney) — If the p-value is lower than 5% the distribution is considered as different between the two treatment groups

66. Secondary Outcome: Change From Baseline in the Dimension 1 Work Productivity and Activity Impairment-Allergy Specific (WPAI-AS) Score: Percentage of Work Time Missed Due to Allergy at Endpoint During the Two-week Treatment Period
Description: The Work Productivity and Activity Impairment-Allergy Specific (WPAI-AS) has been validated to measure generic and allergy-specific performance impairment of work and classroom productivity and of regular daily activity. Higher scores (0% to 100%) indicate greater impairment and a negative change from baseline indicates improvement. Endpoint is defined as the last available postbaseline measurement during the two week treatment period.
Time Frame: Baseline and at endpoint of the 2 week treatment period
Population: Number of participants from the ITT population with available WPAI-AS score (dimension 1) at Endpoint visit and at Baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 225 | 214
percent change | -1.01 (6.76) | -2.68 (11.55)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in WPAI-AS score (dimension 1) at endpoint visit is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.027, ANCOVA — If the p-value of this estimated difference is lower than 5% the mean change from baseline in WPAI-AS score (dimension 1) is considered as different between the two treatment groups; ANCOVA on change from baseline in the WPAI:AS score including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -1.36, 95% CI [-2.56 to -0.16] — The difference presented is 'Levocetirizine 5 mg - Placebo'

67. Secondary Outcome: Change From Baseline in the Dimension 1 Work Productivity and Activity Impairment-Allergy Specific (WPAI-AS) Score: Percentage of Work Time Missed Due to Allergy at Week 1
Description: The Work Productivity and Activity Impairment-Allergy Specific (WPAI-AS) has been validated to measure generic and allergy-specific performance impairment of work and classroom productivity and of regular daily activity. Higher scores (0% to 100%) indicate greater impairment and a negative change from baseline indicates improvement.
Time Frame: Baseline and week 1
Population: Number of participants from the ITT population with available WPAI-AS score (dimension 1) at Week 1 and at Baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 223 | 216
percent change | -1.33 (9.02) | -2.48 (13.79)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in WPAI-AS score (dimension 1) at week 1 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.554, ANCOVA — [p-value comment as in outcome 66, analysis 1]; [statistical method as in outcome 66, analysis 1]; Mean Difference (Final Values) = -0.36, 95% CI [-1.56 to 0.84] — The difference presented is 'Levocetirizine 5 mg - Placebo'

68. Secondary Outcome: Change From Baseline in the Dimension 1 Work Productivity and Activity Impairment-Allergy Specific (WPAI-AS) Score: Percentage of Work Time Missed Due to Allergy at Week 2
Description: as for outcome 67
Time Frame: Baseline and week 2
Population: Number of participants from the ITT population with available WPAI-AS score (dimension 1) at Week 2 and at Baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 218 | 210
percent change | -0.93 (6.78) | -2.83 (11.55)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in WPAI-AS score (dimension 1) at week 2 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.015, ANCOVA — [p-value comment as in outcome 66, analysis 1]; [statistical method as in outcome 66, analysis 1]; Mean Difference (Final Values) = -1.50, 95% CI [-2.72 to -0.29] — The difference presented is 'Levocetirizine 5 mg - Placebo'

69. Secondary Outcome: Change From Baseline in the Dimension 2 Work Productivity and Activity Impairment-Allergy Specific (WPAI-AS) Score: Percentage of Impairment While Working Due to Allergy at Endpoint During the Two-week Treatment Period
Description: as for outcome 66
Time Frame: Baseline and at endpoint of the 2 week treatment period
Population: Number of participants from the ITT population with available WPAI-AS score (dimension 2) at Endpoint visit and at Baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 227 | 216
percent change | -8.06 (23.76) | -13.98 (24.61)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in WPAI-AS score (dimension 2) at endpoint visit is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.016, ANCOVA — If the p-value of this estimated difference is lower than 5% the mean change from baseline in WPAI-AS score (dimension 2) is considered as different between the two treatment groups; [statistical method as in outcome 66, analysis 1]; Mean Difference (Final Values) = -4.60, 95% CI [-8.34 to -0.86] — The difference presented is 'Levocetirizine 5 mg - Placebo'

70. Secondary Outcome: Change From Baseline in the Dimension 2 Work Productivity and Activity Impairment-Allergy Specific (WPAI-AS) Score: Percentage of Impairment While Working Due to Allergy at Week 1
Description: as for outcome 67
Time Frame: Baseline and week 1
Population: Number of participants from the ITT population with available WPAI-AS score (dimension 2) at Week 1 and at Baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 225 | 219
percent change | -5.64 (20.76) | -11.23 (23.04)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in WPAI-AS score (dimension 2) at week 1 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.017, ANCOVA — [p-value comment as in outcome 69, analysis 1]; [statistical method as in outcome 66, analysis 1]; Mean Difference (Final Values) = -4.33, 95% CI [-7.88 to -0.79] — The difference presented is 'Levocetirizine 5 mg - Placebo'

71. Secondary Outcome: Change From Baseline in the Dimension 2 Work Productivity and Activity Impairment-Allergy Specific (WPAI-AS) Score: Percentage of Impairment While Working Due to Allergy at Week 2
Description: as for outcome 67
Time Frame: Baseline and week 2
Population: Number of participants from the ITT population with available WPAI-AS score (dimension 2) at Week 2 and at Baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 220 | 212
percent change | -8.59 (23.57) | -14.34 (24.65)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in WPAI-AS score (dimension 2) at week 2 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.027, ANCOVA — [p-value comment as in outcome 69, analysis 1]; [statistical method as in outcome 66, analysis 1]; Mean Difference (Final Values) = -4.25, 95% CI [-8.02 to -0.47] — The difference presented is 'Levocetirizine 5 mg - Placebo'

72. Secondary Outcome: Change From Baseline in the Dimension 3 Work Productivity and Activity Impairment-Allergy Specific (WPAI-AS) Score: Percentage of Overall Work Impairment Due to Allergy at Endpoint During the Two-week Treatment Period
Description: as for outcome 66
Time Frame: Baseline and at endpoint of the 2 week treatment period
Population: Number of participants from the ITT population with available WPAI-AS score (dimension 3) at Endpoint visit and at Baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 223 | 214
percent change | -8.61 (23.98) | -14.49 (25.43)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in WPAI-AS score (dimension 3) at endpoint visit is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.023, ANCOVA — If the p-value of this estimated difference is lower than 5% the mean change from baseline in WPAI-AS score (dimension 3) is considered as different between the two treatment groups; [statistical method as in outcome 66, analysis 1]; Mean Difference (Final Values) = -4.44, 95% CI [-8.25 to -0.63] — The difference presented is 'Levocetirizine 5 mg - Placebo'

73. Secondary Outcome: Change From Baseline in the Dimension 3 Work Productivity and Activity Impairment-Allergy Specific (WPAI-AS) Score: Percentage of Overall Work Impairment Due to Allergy at Week 1
Description: as for outcome 67
Time Frame: Baseline and week 1
Population: Number of participants from the ITT population with available WPAI-AS score (dimension 3) at Week 1 and at Baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 221 | 216
percent change | -5.80 (20.94) | -11.77 (24.00)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in WPAI-AS score (dimension 3) at week 1 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.015, ANCOVA — [p-value comment as in outcome 72, analysis 1]; [statistical method as in outcome 66, analysis 1]; Mean Difference (Final Values) = -4.56, 95% CI [-8.23 to -0.89] — The difference presented is 'Levocetirizine 5 mg - Placebo'

74. Secondary Outcome: Change From Baseline in the Dimension 3 Work Productivity and Activity Impairment-Allergy Specific (WPAI-AS) Score: Percentage of Overall Work Impairment Due to Allergy at Week 2
Description: as for outcome 67
Time Frame: Baseline and week 2
Population: Number of participants from the ITT population with available WPAI-AS score (dimension 3) at Week 2 and at Baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 216 | 210
percent change | -9.14 (23.78) | -14.89 (25.45)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in WPAI-AS score (dimension 3) at week 2 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.036, ANCOVA — [p-value comment as in outcome 72, analysis 1]; [statistical method as in outcome 66, analysis 1]; Mean Difference (Final Values) = -4.11, 95% CI [-7.95 to -0.27] — The difference presented is 'Levocetirizine 5 mg - Placebo'

75. Secondary Outcome: Change From Baseline in the Dimension 4 Work Productivity and Activity Impairment-Allergy Specific (WPAI-AS) Score: Percentage of Class Time Missed Due to Allergy at Endpoint During the Two-week Treatment Period
Description: as for outcome 66
Time Frame: Baseline and at endpoint of the 2 week treatment period
Population: Number of participants from the ITT population with available WPAI-AS score (dimension 4) at Endpoint visit and at Baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 30 | 22
percent change | 0.25 (11.50) | -3.64 (12.84)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in WPAI-AS score (dimension 4) at endpoint visit is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.102, ANCOVA — If the p-value of this estimated difference is lower than 5% the mean change from baseline in WPAI-AS score (dimension 4) is considered as different between the two treatment groups; [statistical method as in outcome 66, analysis 1]; Mean Difference (Final Values) = -4.51, 95% CI [-9.95 to 0.93] — The difference presented is 'Levocetirizine 5 mg - Placebo'

76. Secondary Outcome: Change From Baseline in the Dimension 4 Work Productivity and Activity Impairment-Allergy Specific (WPAI-AS) Score: Percentage of Class Time Missed Due to Allergy at Week 1
Description: as for outcome 67
Time Frame: Baseline and week 1
Population: Number of participants from the ITT population with available WPAI-AS score (dimension 4) at Week 1 and at Baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 27 | 24
percent change | -2.82 (9.16) | -3.27 (14.04)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in WPAI-AS score (dimension 4) at week 1 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.493, ANCOVA — [p-value comment as in outcome 75, analysis 1]; [statistical method as in outcome 66, analysis 1]; Mean Difference (Final Values) = -1.44, 95% CI [-5.66 to 2.78] — The difference presented is 'Levocetirizine 5 mg - Placebo'

77. Secondary Outcome: Change From Baseline in the Dimension 4 Work Productivity and Activity Impairment-Allergy Specific (WPAI-AS) Score: Percentage of Class Time Missed Due to Allergy at Week 2
Description: as for outcome 67
Time Frame: Baseline and week 2
Population: Number of participants from the ITT population with available WPAI-AS score (dimension 4) at Week 2 and at Baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 29 | 22
percent change | -0.03 (11.60) | -3.64 (12.84)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in WPAI-AS score (dimension 4) at week 2 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.117, ANCOVA — [p-value comment as in outcome 75, analysis 1]; [statistical method as in outcome 66, analysis 1]; Mean Difference (Final Values) = -4.38, 95% CI [-9.91 to 1.15] — The difference presented is 'Levocetirizine 5 mg - Placebo'

78. Secondary Outcome: Change From Baseline in the Dimension 5 Work Productivity and Activity Impairment-Allergy Specific (WPAI-AS) Score: Percentage of Impairment in the Classroom Due to Allergy at Endpoint During the Two-week Treatment Period
Description: as for outcome 66
Time Frame: Baseline and at endpoint of the 2 week treatment period
Population: Number of participants from the ITT population with available WPAI-AS score (dimension 5) at Endpoint visit and at Baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 30 | 22
percent change | -6.33 (22.05) | -7.73 (24.09)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in WPAI-AS score (dimension 5) at endpoint visit is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.409, ANCOVA — If the p-value of this estimated difference is lower than 5% the mean change from baseline in WPAI-AS score (dimension 5) is considered as different between the two treatment groups; [statistical method as in outcome 66, analysis 1]; Mean Difference (Final Values) = -4.58, 95% CI [-15.65 to 6.49] — The difference presented is 'Levocetirizine 5 mg - Placebo'

79. Secondary Outcome: Change From Baseline in the Dimension 5 Work Productivity and Activity Impairment-Allergy Specific (WPAI-AS) Score: Percentage of Impairment in the Classroom Due to Allergy at Week 1
Description: as for outcome 67
Time Frame: Baseline and week 1
Population: Number of participants from the ITT population with available WPAI-AS score (dimension 5) at Week 1 and at Baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 28 | 25
percent change | -2.86 (23.70) | -6.00 (24.66)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in WPAI-AS score (dimension 5) at week 1 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.432, ANCOVA — [p-value comment as in outcome 78, analysis 1]; [statistical method as in outcome 66, analysis 1]; Mean Difference (Final Values) = -4.54, 95% CI [-16.10 to 7.01] — The difference presented is 'Levocetirizine 5 mg - Placebo'

80. Secondary Outcome: Change From Baseline in the Dimension 5 Work Productivity and Activity Impairment-Allergy Specific (WPAI-AS) Score: Percentage of Impairment in the Classroom Due to Allergy at Week 2
Description: as for outcome 67
Time Frame: Baseline and week 2
Population: Number of participants from the ITT population with available WPAI-AS score (dimension 5) at Week 2 and at Baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 29 | 22
percent change | -6.55 (22.40) | -7.73 (24.09)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in WPAI-AS score (dimension 5) at week 2 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.450, ANCOVA — [p-value comment as in outcome 78, analysis 1]; [statistical method as in outcome 66, analysis 1]; Median Difference (Final Values) = -4.24, 95% CI [-15.46 to 6.99] — The difference presented is 'Levocetirizine 5 mg - Placebo'

81. Secondary Outcome: Change From Baseline in the Dimension 6 Work Productivity and Activity Impairment-Allergy Specific (WPAI-AS) Score: Percentage of Overall Classroom Impairment Due to Allergy at Endpoint During the Two-week Treatment Period
Description: as for outcome 66
Time Frame: Baseline and at endpoint of the 2 week treatment period
Population: Number of participants from the ITT population with available WPAI-AS score (dimension 6) at Endpoint visit and at Baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 30 | 22
percent change | -5.22 (21.53) | -8.65 (24.78)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in WPAI-AS score (dimension 6) at endpoint visit is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.251, ANCOVA — If the p-value of this estimated difference is lower than 5% the mean change from baseline in WPAI-AS score (dimension 6) is considered as different between the two treatment groups; [statistical method as in outcome 66, analysis 1]; Mean Difference (Final Values) = -6.37, 95% CI [-17.40 to 4.67] — The difference presented is 'Levocetirizine 5 mg - Placebo'

82. Secondary Outcome: Change From Baseline in the Dimension 6 Work Productivity and Activity Impairment-Allergy Specific (WPAI-AS) Score: Percentage of Overall Classroom Impairment Due to Allergy at Week 1
Description: as for outcome 67
Time Frame: Baseline and week 1
Population: Number of participants from the ITT population with available WPAI-AS score (dimension 6) at Week 1 and at Baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 27 | 24
percent change | -3.05 (24.92) | -7.18 (26.96)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in WPAI-AS score (dimension 6) at week 1 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.258, ANCOVA — [p-value comment as in outcome 81, analysis 1]; [statistical method as in outcome 66, analysis 1]; Mean Difference (Final Values) = -7.06, 95% CI [-19.48 to 5.36] — The difference presented is 'Levocetirizine 5 mg - Placebo'

83. Secondary Outcome: Change From Baseline in the Dimension 6 Work Productivity and Activity Impairment-Allergy Specific (WPAI-AS) Score: Percentage of Overall Classroom Impairment Due to Allergy at Week 2
Description: as for outcome 67
Time Frame: Baseline and week 2
Population: Number of participants from the ITT population with available WPAI-AS score (dimension 6) at Week 2 and at Baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 29 | 22
percent change | -5.52 (21.85) | -8.65 (24.78)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in WPAI-AS score (dimension 6) at week 2 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.288, ANCOVA — [p-value comment as in outcome 81, analysis 1]; [statistical method as in outcome 66, analysis 1]; Mean Difference (Final Values) = -5.96, 95% CI [-17.13 to 5.22] — The difference presented is 'Levocetirizine 5 mg - Placebo'

84. Secondary Outcome: Change From Baseline in the Dimension 7 Work Productivity and Activity Impairment-Allergy Specific (WPAI-AS) Score: Percentage of Activity Impairment Due to Allergy at Endpoint During the Two-week Treatment Period
Description: as for outcome 66
Time Frame: Baseline and at endpoint of the 2 week treatment period
Population: Number of participants from the ITT population with available WPAI-AS score (dimension 7) at Endpoint visit and at Baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 280 | 273
percent change | -11.71 (23.40) | -18.46 (24.43)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in WPAI-AS score (dimension 7) at endpoint visit is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — If the p-value of this estimated difference is lower than 5% the mean change from baseline in WPAI-AS score (dimension 7) is considered as different between the two treatment groups; [statistical method as in outcome 66, analysis 1]; Mean Difference (Final Values) = -5.91, 95% CI [-9.34 to -2.47] — The difference presented is 'Levocetirizine 5 mg - Placebo'

85. Secondary Outcome: Change From Baseline in the Dimension 7 Work Productivity and Activity Impairment-Allergy Specific (WPAI-AS) Score: Percentage of Activity Impairment Due to Allergy at Week 1
Description: as for outcome 67
Time Frame: Baseline and week 1
Population: Number of participants from the ITT population with available WPAI-AS score (dimension 7) at Week 1 and at Baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 279 | 273
percent change | -6.85 (19.69) | -14.29 (23.32)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in WPAI-AS score (dimension 7) at week 1 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p < 0.001, ANCOVA — [p-value comment as in outcome 84, analysis 1]; [statistical method as in outcome 66, analysis 1]; Mean Difference (Final Values) = -6.62, 95% CI [-9.88 to -3.35] — The difference presented is 'Levocetirizine 5 mg - Placebo'

86. Secondary Outcome: Change From Baseline in the Dimension 7 Work Productivity and Activity Impairment-Allergy Specific (WPAI-AS) Score: Percentage of Activity Impairment Due to Allergy at Week 2
Description: as for outcome 67
Time Frame: Baseline and week 2
Population: Number of participants from the ITT population with available WPAI-AS score (dimension 7) at Week 2 and at Baseline
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 273 | 267
percent change | -12.05 (23.53) | -18.84 (24.43)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in WPAI-AS score (dimension 7) at week 2 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.001, ANCOVA — [p-value comment as in outcome 84, analysis 1]; [statistical method as in outcome 66, analysis 1]; Mean Difference (Final Values) = -5.69, 95% CI [-9.16 to -2.21] — The difference presented is 'Levocetirizine 5 mg - Placebo'

87. Secondary Outcome: Change From Baseline in Epworth Sleepiness Scale (ESS) Score at Endpoint During the Two-week Treatment Period
Description: The Epworth Sleepiness Scale (ESS) is the criterion standard for measuring daytime sleepiness in adults. Subjects are asked to rate the chances of dozing off or falling asleep in eight situations encountered in daily life on a scale of 0 to 3, with scores ranging from 0 to 24. A score >= 8 indicates sleepiness. Endpoint is defined as the last available postbaseline measurement during the two week treatment period.
Time Frame: Baseline and at endpoint of the 2 week treatment period
Population: Number of participants from the ITT population with available ESS score at Endpoint visit and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 284
points on a scale | -1.02 (3.84) | -1.79 (4.16)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in ESS score at endpoint visit is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.027, ANCOVA — If the p-value of this estimated difference is lower than 5% the mean change from baseline in ESS score is considered as different between the two treatment groups; ANCOVA on change from baseline in ESS score including treatment and pooled center as factors and baseline mean score as covariate; Mean Difference (Final Values) = -0.68, 95% CI [-1.29 to -0.08] — The difference presented is 'Levocetirizine 5 mg - Placebo'

88. Secondary Outcome: Change From Baseline in Epworth Sleepiness Scale (ESS) Score at Week 1
Description: The Epworth Sleepiness Scale (ESS) is the criterion standard for measuring daytime sleepiness in adults. Subjects are asked to rate the chances of dozing off or falling asleep in eight situations encountered in daily life on a scale of 0 to 3, with scores ranging from 0 to 24. A score >= 8 indicates sleepiness.
Time Frame: Baseline and week 1
Population: Number of participants from the ITT population with available ESS score at Week 1 and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 288 | 280
points on a scale | -0.67 (3.33) | -0.91 (3.65)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in ESS score at week 1 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.535, ANCOVA — [p-value comment as in outcome 87, analysis 1]; [statistical method as in outcome 87, analysis 1]; Mean Difference (Final Values) = -0.17, 95% CI [-0.70 to 0.37] — The difference presented is 'Levocetirizine 5 mg - Placebo'

89. Secondary Outcome: Change From Baseline in Epworth Sleepiness Scale (ESS) Score at Week 2
Description: as for outcome 88
Time Frame: Baseline and week 2
Population: Number of participants from the ITT population with available ESS score at Week 2 and at Baseline
Measure: Mean (Standard Deviation); unit: points on a scale
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 286 | 278
points on a scale | -1.05 (3.88) | -1.78 (4.20)
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The mean change from baseline in ESS score at week 2 is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.042, ANCOVA — [p-value comment as in outcome 87, analysis 1]; [statistical method as in outcome 87, analysis 1]; Mean Difference (Final Values) = -0.64, 95% CI [-1.26 to -0.02] — The difference presented is 'Levocetirizine 5 mg - Placebo'

90. Secondary Outcome: Sleepiness According to Epworth Sleepiness Scale (ESS) Score at Baseline and at Endpoint During the Two-week Treatment Period
Description: as for outcome 87
Time Frame: Baseline and at endpoint of the 2 week treatment period
Population: Number of participants from the ITT population
Measure: Number; unit: participants
Arm/Group | Placebo | Levocetirizine
Number analyzed (Participants) | 293 | 287
participants
  ESS score < 8 at Baseline and < 8 at Endpoint | 66 | 63
  ESS score < 8 at Baseline and ≥ 8 at Endpoint | 16 | 13
  ESS score ≥ 8 at Baseline and < 8 at Endpoint | 46 | 57
  ESS score ≥ 8 at Baseline and ≥ 8 at Endpoint | 165 | 151
Statistical Analysis 1: Comparison: Placebo vs Levocetirizine; The Null Hypothesis is expressed as follows: 'The change from baseline to endpoint visit in score category (ESS score < 8 or >= 8) is not different from subjects treated with levocetirizine than subjects treated with placebo.'; Test type: Superiority or Other; p = 0.171, Repeated measure analysis (CATMOD) — If the p-value of this estimated difference is lower than 5% the change from baseline is considered as different between the two treatment groups

ADVERSE EVENTS:
Time Frame: 14 days
Description: Safety population consists of all randomized subjects treated at least once during two week treatment period (578 subjects).
Arm/Group | Placebo | Levocetirizine
Serious Adverse Events (participants affected / at risk) | 0/293 | 1/285
Other Adverse Events (participants affected / at risk) | 12/293 | 13/285
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=293) | Levocetirizine (N=285)
Cellulitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=293) | Levocetirizine (N=285)
Headache (Nervous system disorders) | 12 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
UCB has > 60 days but <= 180 days to review results communications prior to public release and may delete information that compromises ongoing studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.